CLINICAL TRIAL: NCT02713243
Title: A Double Blind, Randomized Placebo Controlled Crossover Multiple Dose Study of LJN452 to Assess Safety, Tolerability and Efficacy in Patients With Primary Bile Acid Diarrhea (pBAD).
Brief Title: To Assess Safety, Tolerability and Efficacy of LJN452 in Patients With Primary Bile Acid Diarrhea.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLJN452X2202; 2015-003192-30 (EudraCT Number)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-08

CONDITIONS: Primary Bile Acid Diarrhea
Keywords: Primary bile acid diarrhea,; FXR agonist,; bile acid malabsorption.
MeSH Terms: interventions — tropifexor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LJN452 followed by placebo (Experimental): Randomized patients in this arm will receive single oral dose of LJN452 daily for 14 days. There will be a washout period between 7 to 28 days followed by single oral dose of placebo daily for 14 days.
  Interventions: Drug: LJN452; Drug: Placebo to LJN452
- Placebo followed by LJN452 (Experimental): Randomized patients in this arm will receive single oral dose of placebo daily for 14 days. There will be a washout period between 7 to 28 days followed by single oral dose of LJN452 daily for 14 days.
  Interventions: Drug: LJN452; Drug: Placebo to LJN452

INTERVENTIONS:
Drug: LJN452 — Capsules containing LJN452
Drug: Placebo to LJN452 — Capsules containing placebo to LJN452

SUMMARY:
The purpose of this study is to determine whether LJN452 improves the symptoms of bile acid diarrhea and to assess its safety and tolerability profile in patients with primary bile acid diarrhea (pBAD) to guide decision-making regarding further clinical development in this indication.

ELIGIBILITY:
Key Inclusion Criteria:

* A history of diarrheal symptoms for at least 3 months prior to dosing - Average stool frequency of at least 2 per day when off therapy AND Average stool form of >5 on Bristol Stool Chart.
* Previous laboratory or radiological confirmation of bile acid malabsorption with either fecal bile acid loss OR 7 day 75Selenium homocholic acid taurine (75SeHCAT) retention.
* Age ≥ 18 years.

Key Exclusion Criteria:

* Patients with other diagnoses leading to diarrhea, including colorectal neoplasia, ulcerative colitis, Crohn's disease, celiac disease, chronic pancreatitis, drug-induced diarrhea or active infection AND Patients who have not been investigated by standard clinical assessments to exclude these disorders.
* Treatment with bile acid sequestrants (colestyramine, colestipol, colesevelam) for 2 weeks before the first dose of LJN452. A washout of 14 days for these agents will be allowed before first dosing.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* A positive Hepatitis B surface antigen or Hepatitis C test result.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Rochester, Minnesota, United States
- United Kingdom (3):
  - Novartis Investigative Site, Harrow, Middlesex
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield

REFERENCES:
- [Derived] Camilleri M, Nord SL, Burton D, Oduyebo I, Zhang Y, Chen J, Im K, Bhad P, Badman MK, Sanders DS, Walters JRF. Randomised clinical trial: significant biochemical and colonic transit effects of the farnesoid X receptor agonist tropifexor in patients with primary bile acid diarrhoea. Aliment Pharmacol Ther. 2020 Sep;52(5):808-820. doi: 10.1111/apt.15967. Epub 2020 Jul 23. PMID 32702169
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 20 patients were enrolled in this study and received at least one dose of LJN452 or matching placebo for 14 days in Period 1. There will be a washout period between 7 to 28 days followed by Period 2 drug if patient on LJN452 or Placebo in Period 1 they will take Placebo or LJN452 respectively in Period 2 for 14 days
Period: Overall Study
Arm/Group | LJN452 Followed by Placebo | Placebo Followed by LJN452
Started | 10 | 10
PD Analysis Set | 9 | 10
PK Analysis Set | 8 | 9
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Abnormal laboratory value(s)# | 1 | 0
Not completed — Administrative problems | 0 | 1
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LJN452 Followed by Placebo | Placebo Followed by LJN452 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.25) | 57.9 (16.47) | 53.7 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reported With Adverse Events , Serious Adverse Events and Death.
Description: Number of patients reported with adverse events , serious adverse events and death.
Time Frame: up to Day 79
Population: Safety analysis set consists of 20 patients(10 pts per treatment period),17 &19 patients received at least 1 LJN & 1 Placebo dose, respectively, therefore 17 pts in the LJN452 &19 in the Placebo treatment periods were analyzed. Adverse events were summarized using descriptive statistics only with no formal statistical analysis performed.
Measure: Number; unit: count of participants
Groups:
- LJN452 ALL Patients: All Patients on LJN452 in both Period 1 and Period 2
- Placebo ALL Patients: All Patients on Placebo in both Period 1 and Period 2
Arm/Group | LJN452 ALL Patients | Placebo ALL Patients
Number analyzed (Participants) | 17 | 19
count of participants
  AEs, Patients with AEs | 9 | 14
  Study drug-related AEs | 0 | 4
  Serious AEs | 0 | 0
  Death | 0 | 0

2. Primary Outcome: Stool Frequency at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 Combined
Description: Stool frequency at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 combined
Time Frame: Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 combined
Population: PD analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Stools per week
Arm/Group | LJN452 ALL Patients | Placebo ALL Patients
Number analyzed (Participants) | 20 | 20
Stools per week
  Baseline: number analyzed (Participants) | 15 | 18
  Baseline | 18.0 (9.39) | 15.9 (6.92)
  Week 1 (Period 1 & 2): number analyzed (Participants) | 16 | 18
  Week 1 (Period 1 & 2) | 20.0 (11.62) | 16.2 (7.19)
  Week 2 (Period 1 & 2): number analyzed (Participants) | 15 | 18
  Week 2 (Period 1 & 2) | 18.8 (9.68) | 17.5 (10.88)
  Week 1 & 2(Period 1 & 2) | 19.4 (10.56) | 16.8 (9.11)
Statistical Analysis 1: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 1 (Period 1 & 2); Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Net) = 4.04, 95% CI 2-sided [0.98 to 7.11]
Statistical Analysis 2: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 2 (Period 1 & 2); Test type: Superiority; p = 0.401, Mixed Models Analysis; Mean Difference (Net) = 1.31, 95% CI 2-sided [-1.77 to 4.38]
Statistical Analysis 3: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 1&2 (Period 1 & 2); Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Net) = 2.67, 95% CI 2-sided [0.46 to 4.89]

3. Secondary Outcome: Area Under the Plasma Concentration-time Profile (AUCtau) of LJN452
Description: AUCtau- is the area under the plasma (or serum or blood) concentration-time curve from time zero to the end of the dosing interval tau [mass x time / volume]
Time Frame: Day 1 (Period 1 & 2) and Day 12 (Period 1 & 2)
Population: PK analysis set: Patients with at least one valid PK concentration measurement and no major protocol deviations affecting PK No statistical Analysis
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LJN452 ALL Patients
Number analyzed (Participants) | 17
hr*ng/mL
  Day 1: number analyzed (Participants) | 7
  Day 1 | 23.6 (7.24)
  Day 12: number analyzed (Participants) | 5
  Day 12 | 22.1 (4.83)

4. Secondary Outcome: (Cmax) of LJN452
Description: Cmax is the observed maximum plasma (or serum or blood) concentration following drug administration [mass / volume]
Time Frame: Day 1 (Period 1 & 2) and Day 12 (Period 1 & 2)
Population: PK analysis set: Patients with at least one valid PK concentration measurement and no major protocol deviations affecting PK - No statistical Analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LJN452 ALL Patients
Number analyzed (Participants) | 17
ng/mL
  Day 1: number analyzed (Participants) | 9
  Day 1 | 1.63 (0.414)
  Day 12: number analyzed (Participants) | 15
  Day 12 | 1.82 (0.704)

5. Secondary Outcome: Time to Reach Maximum Concentration After Drug Administration (Tmax)
Description: Tmax is the time to reach the maximum concentration after drug administration [time]
Time Frame: Day 1 (Period 1 & 2) and Day 12 (Period 1 & 2)
Population: PK analysis set: Patients with at least one valid PK concentration measurement and no major protocol deviations affecting PK; No statistical Analysis
Measure: Median (Full Range); unit: hr
Arm/Group | LJN452 ALL Patients
Number analyzed (Participants) | 17
hr
  Day 1: number analyzed (Participants) | 9
  Day 1 | 5.00 [3.92 to 8.00]
  Day 12: number analyzed (Participants) | 15
  Day 12 | 5.00 [1.83 to 8.00]

6. Secondary Outcome: Total Dose of Rescue Medication Used at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 Combined
Description: Total Dose of Rescue Medication used at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 combined; Rescue Medication used was loperamide
Time Frame: Baseline, Week 1 (Period 1 & 2), Week 2 (Period 1 & 2), Week 1 & 2 combined
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | LJN452 ALL Patients | Placebo ALL Patients
Number analyzed (Participants) | 20 | 20
mg
  Baseline: number analyzed (Participants) | 16 | 18
  Baseline | 0.9 (3.50) | 1.3 (5.66)
  Week 1 (Period 1 & 2): number analyzed (Participants) | 16 | 18
  Week 1 (Period 1 & 2) | 0.6 (1.75) | 0.7 (2.06)
  Week 2 (Period 1 & 2): number analyzed (Participants) | 16 | 18
  Week 2 (Period 1 & 2) | 0.5 (1.37) | 0.7 (1.68)
  Week 1 & 2(Period 1 & 2) | 0.6 (1.54) | 0.7 (1.85)

7. Primary Outcome: Stool Form at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 Combined
Description: Stool Form at Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 combined Clinical Symptoms will be measured as change from baseline in stool types per Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify feces on a scale from 1 to 7 according to increasing wateriness.
Time Frame: Baseline, Week 1 (Period 1 & Period 2), Week 2 (Period 1 & Period 2), and Week 1 & 2 combined
Population: PD analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LJN452 ALL Patients | Placebo ALL Patients
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline: number analyzed (Participants) | 15 | 18
  Baseline | 5.5 (0.87) | 5.1 (0.94)
  Week 1 (Period 1 & 2): number analyzed (Participants) | 16 | 18
  Week 1 (Period 1 & 2) | 5.3 (0.78) | 5.3 (0.79)
  Week 2 (Period 1 & 2): number analyzed (Participants) | 15 | 18
  Week 2 (Period 1 & 2) | 4.9 (0.82) | 5.1 (1.01)
  Week 1 & 2(Period 1 & 2) | 5.1 (0.81) | 5.2 (0.90)
Statistical Analysis 1: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 1 (Period 1 & 2); Test type: Superiority; p = 0.533, Mixed Models Analysis; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.27 to 0.52]
Statistical Analysis 2: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 2 (Period 1 & 2); Test type: Superiority; p = 0.640, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.49 to 0.30]
Statistical Analysis 3: Comparison: LJN452 ALL Patients vs Placebo ALL Patients; Week 1&2 (Period 1 & 2); Test type: Superiority; p = 0.916, Mixed Models Analysis; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.27 to 0.30]

ADVERSE EVENTS:
Time Frame: Adverse Events are monitored from date of First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) Day 79. All other adverse events are monitored from First Patient First Treatment until Last Patient Last Visit (Day 79).
Description: Safety analysis set consists of 20 patients(10 pts per treatment period),17 &19 patients received at least 1 LJN & 1 Placebo dose, respectively, therefore 17 pts in the LJN452 &19 in the Placebo treatment periods were analyzed. Adverse events were summarized using descriptive statistics only with no formal statistical analysis performed.
Arm/Group | LJN452 ALL Patients | Placebo ALL Patients
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 9/17 | 14/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 ALL Patients (N=17) | Placebo ALL Patients (N=19)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Bile acid malabsorption (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Biliary dyspepsia (Hepatobiliary disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 4
Migraine (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02713243/SAP_001.pdf
  • Study Protocol (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02713243/Prot_002.pdf